CLINICAL TRIAL: NCT00186641
Title: High Dose Chemotherapy and Peripheral Blood Progenitor Cell Rescue for Patients With Breast Cancer
Brief Title: High Dose Chemotherapy and Autologous Transplant for Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stanford University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT42
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2007-07-11 (Estimated); Status verified 2007-07

CONDITIONS: Graft vs Host Disease
Keywords: chronic Graft vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Drug Therapy

INTERVENTIONS:
Procedure: high dose chemo and auto hematopoietic cell transplant

SUMMARY:
To determine survival outcomes for patients with chemosensitive brest cancer after treatment with high dose chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Stage II, III or IV breast cancer
* chemosensitive
* adequate organ function

Exclusion Criteria:

* prior transplant,
* life threatening disease
* brain metastases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Study Completion 2005-03

PRIMARY OUTCOMES:
Survival

CONTACTS AND LOCATIONS:
Overall Officials: Ginna Laport, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Cancer Center, Stanford, California, United States